CLINICAL TRIAL: NCT00723567
Title: Case Report: A Novel Mutation of the Spectrin Gene in a Family of Northern European Descent Is Associated With Three Different Phenotypes
Brief Title: A Novel Mutation of the Spectrin Gene
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: University of Witwatersrand, South Africa (Other)
Responsible Party: Josef T. Prchal, MD, University of Utah
Other Study IDs: 27669
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Hereditary Elliptocytosis (HE); Hereditary Pyropoikilocytosis (HPP)
Keywords: Spectrin Gene; Hereditary Elliptocytosis (HE); Hereditary Pyropoikilocytosis (HPP); Genetics
MeSH Terms: conditions — Elliptocytosis, Hereditary; Pyropoikilocytosis, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Affected Group: Family members of northern European descent in which members have different erythrocyte morphology ranging from atypical HPP to HE to normal and a novel Sp mutation.

SUMMARY:
The purpose of this study is to find a gene or its mutation (an altered gene) that puts individuals at risk for developing HE or HPP.

DETAILED DESCRIPTION:
Mutations of spectrin (Sp) involving the Sp heterodimer self-association site (the I domain of Sp) represent the most common group of membrane skeletal defects in hereditary elliptocytosis (HE) and a closely related disorder, hereditary pyropoikilocytosis (HPP). HPP is characterized by extreme anisocytic microcytosis, a severe spectrin dimer self-association defect and spectrin deficiency. The conventional explanation for the different phenotypes is that HPP subjects are compound heterozygotes for an sp defect that interferes with sp tetramer assembly and a second defect which results in decreased synthesis of functional sp. In contrast, HE subjects have normal spectrin content and a less severe sp self-association defect. The clinical expression of HE/HPP is influenced by the inheritance of modifying factors such as the Sp hypomorphic mutation, LELY. LELY is a low expression allele of the Sp gene characterized by a C>G mutation in codon 1857 of exon 40 and a C>T -12 mutation in intron 45 that is responsible for partial skipping of exon 46, which is essential for the functional assembly of /b sp dimers.

CASE REPORT:

Here we describe four members from a family of northern European descent in which members had different erythrocyte morphology ranging from atypical HPP to HE to normal and a novel Sp mutation. Quantitation of RBC membrane proteins of the propositus with atypical non-microcytic HPP revealed 48% spectrin dimers (control 10%) due to a marked increase in the 74kD I Sp peptide. There was only a slight decrease in the spectrin/band 3 ratio, which correlated with the normocytic morphology. There was also an abnormal Sp peptide at 41kD suggesting presence of LELY. Sequencing of his Sp gene revealed heterozygosity for a novel mutation in exon 2, codon 34: CGG->CCG (Arg>Pro) and heterozygosity for LELY. These mutations were also present in his brother and daughter who have HE, while another son, who had Arg34Pro, but not LELY has repeatedly confirmed normal morphology.

We plan to screen 11 other family members who are suspected to have HPP or HE. Blood samples will be obtained and the following will be performed:

1. Quantitation of erythrocyte (RBC) membrane proteins
2. DNA extraction from the WBC and screening for spectrin mutation with restriction enzymes (if needed we will sequence spectrin gene)
3. Quantitative Real Time PCR testing will be done on RNA to assess the spectrin gene expression
4. History, Clinical examination, CBC, chemistry and peripheral blood smear

Quantitation of RBC membrane proteins will be done by looking for the abnormal increase in the amount of spectrin dimers in patients with HPP (control 10%). We will also look at the DNA for any known or yet unreported mutations in the spectrin gene and we will correlate the expression of spectrin gene wrt level of spectrin protein in the RNA.

No statistical analysis will be done. This is an observation study designed to correlate clinical features with the above mentioned tests results.

ELIGIBILITY:
Inclusion Criteria:

* > 7 years of age
* Consenting family members

Exclusion Criteria:

* Anyone not meeting the criteria above

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Members from a family of northern European descent in which members had different erythrocyte morphology ranging from atypical HPP to HE to normal and a novel Sp mutation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Identify a gene or its mutation (an altered gene) that puts individuals at risk for developing HE or HPP | After sample is obtained

CONTACTS AND LOCATIONS:
Overall Officials: Josef T Prchal, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Ivanov IT, Tolekova A, Chakaarova P. Erythrocyte membrane defects in hemolytic anemias found through derivative thermal analysis of electric impedance. J Biochem Biophys Methods. 2007 Jun 10;70(4):641-8. doi: 10.1016/j.jbbm.2007.02.004. Epub 2007 Mar 1. PMID 17395266
- [Background] Ramos MC, Schafernak KT, Peterson LC. Hereditary pyropoikilocytosis: a rare but potentially severe form of congenital hemolytic anemia. J Pediatr Hematol Oncol. 2007 Feb;29(2):128-9. doi: 10.1097/MPH.0b013e3180320b6f. PMID 17279012
- [Background] King MJ, Telfer P, MacKinnon H, Langabeer L, McMahon C, Darbyshire P, Dhermy D. Using the eosin-5-maleimide binding test in the differential diagnosis of hereditary spherocytosis and hereditary pyropoikilocytosis. Cytometry B Clin Cytom. 2008 Jul;74(4):244-50. doi: 10.1002/cyto.b.20413. PMID 18454487
- [Background] An X, Mohandas N. Disorders of red cell membrane. Br J Haematol. 2008 May;141(3):367-75. doi: 10.1111/j.1365-2141.2008.07091.x. Epub 2008 Mar 12. PMID 18341630
- [Background] Gaetani M, Mootien S, Harper S, Gallagher PG, Speicher DW. Structural and functional effects of hereditary hemolytic anemia-associated point mutations in the alpha spectrin tetramer site. Blood. 2008 Jun 15;111(12):5712-20. doi: 10.1182/blood-2007-11-122457. Epub 2008 Jan 24. PMID 18218854
- [Background] Salomao M, Zhang X, Yang Y, Lee S, Hartwig JH, Chasis JA, Mohandas N, An X. Protein 4.1R-dependent multiprotein complex: new insights into the structural organization of the red blood cell membrane. Proc Natl Acad Sci U S A. 2008 Jun 10;105(23):8026-31. doi: 10.1073/pnas.0803225105. Epub 2008 Jun 4. PMID 18524950